## "USEFULNESS OF VIRTUAL REALITY IN THE MANAGEMENT OF PAIN ASSOCIATED WITH VENIPUNCTURE IN PEDIATRICS: A MULTICENTER RANDOMIZED CLINICAL TRIAL (RealPED)" ANNEX 1: PATIENT INFORMATION SHEET AND INFORMED CONSENT

Date: December 22, 2021

The Pediatrics Service of the Xàtiva-Ontinyent Health Department is carrying out a research project entitled: "USEFULNESS OF VIRTUAL REALITY IN THE MANAGEMENT OF PAIN ASSOCIATED WITH VENIPUNCTURE IN PEDIATRICS: A MULTICENTER RANDOMIZED CLINICAL TRIAL (RealPED)".

This study aims to test whether the use of virtual reality during a blood test reduces the pain and anxiety associated with such extraction. After accepting participation in the study, each child will be randomly assigned to 2 groups: one with virtual reality and one with usual care.

No adverse effects are expected to appear since the use of virtual reality glasses is controlled and for a limited time (only during blood test), but headaches and dizziness have been described in some patients.

| After knowing this information: I, | . (name and surname) |
|---|---|
| ask questions about the study. I have | formation sheet given to me. I have been able to received enough information and I have been data confidentially following the legal regulations ction of Personal Data). |
| I have spoken to: | (name of the collaborating researcher). |
| · | udy is voluntary, and that I can withdraw from xplanations and without affecting the medical eely agree. |
| Signature and date: | |
| Mother / father / legal tutor | Collaborating Researcher |